CLINICAL TRIAL: NCT04155177
Title: Learning Curve of the "French Ambulatory Caesarean Section"
Brief Title: FAUCS Surgery: Learning Curve for Resident
Status: Withdrawn | Type: Observational
Why Stopped: no participants because of the sars cov 2 pandemic there is no volonteer to be recruited for the lurning curve . all the residents are busy working in COVID UNITS
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaouther Dimassi, Associate professor, University Tunis El Manar
Other Study IDs: 36211361
Record Dates: First submitted 2019-10-15; First posted 2019-11-07 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Caesarean; Training
Keywords: Caesarean; surgery; training; obstetrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- begining of curriculum: trainees in obstetrics and gynecology who have achieved less than 2 years of their hole curriculum
  Interventions: Procedure: training for french ambulatory caesarean section
- mid curriculum: trainees in obstetrics and gynecology who have achieved at least 2 years and less than 4 years of their hole curriculum
  Interventions: Procedure: training for french ambulatory caesarean section
- Advanced: trainees in obstetrics and gynecology who have achieved at least 4 years of their hole curriculm
  Interventions: Procedure: training for french ambulatory caesarean section

INTERVENTIONS:
Procedure: training for french ambulatory caesarean section — The participant will be first invited to consult a theoretical support and a video treating on FAUCS.
  After that, he will be asked to be the first assistant, in a FAUCS procedure with one of the two senior surgeons assigned for the study.
  In a second step, the trainee will have to perform all the steps of the FAUCS, assisted by one of the two senior surgeons . During each surgery, Operative time will be measured, while an evaluation on four stages according to the Zwisch model of supervision will performed by the senior surgeons .
  Once, the two seniors agree on the highest level assessment for the resident, he will be allowed to operate alone FAUCS procedures and will be evaluated by the measurement of operating times, the neonatal outcomes and the occurrence or not of complications.
  finally, total number of FAUCS procedures required for each resident in order to master the technique will be determined.

SUMMARY:
In the last decades, caesarean section (CS) rates are getting higher in all over the world.

This encourages us to improve operative techniques. In January 2018, investigators have introduced in the study unit: The French Ambulatory C section (FAUCS). This innovative approach appeares to provide a shorter recovery time, with a hospital discharge the day after surgery in 90% and then a better experience of childbirth.

The diffusion of this technique requires its integration to the curriculum of residency.

In this study, investigators will determine the mean number of procedures needed for trainees to master FAUCS.

DETAILED DESCRIPTION:
Caesarean section (CS) is of the most commonly performed operations worldwide. This encourages a permanent search to improve the operative techniques for a better childbirth experience. The MisgavLadach (MLC), caesarean section is the gold standard for caesarean section. Thus so, it is included During the first years of obstetrics curriculum.

In January 2018, investigators have introduced The French Ambulatory C section (FAUCS) in the study unit. It is an innovative approach for CS. combining a left paramedian incision , an extra peritoneal access to the uterus and a purse-string double-layer closure of the uterus. Since that date, two doctors practice it regularly. However, the diffusion of this technique requires its integration into the curriculum of residency. Currently, there is no study on the learning procedure of FAUCS.

In our study, investigators will determine the mean number of procedures needed for trainees to master FAUCS.

Once the resident will master the procedure, investigators will study his skills evolution every 5 surgeries performed alone.

ELIGIBILITY:
Inclusion Criteria:

* trainee in obstetrics and gynecology.
* trainee subscribed for a training programm in the suty unit during the study period

Exclusion Criteria :

* Trainee in obstetrics and gynecology subscribed in atraining program elswhere from the sutudy unit during the study period
* trainee who refused to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all the included participants will be enrolled in three groups :
  * First group : trainees in obstetrics and gynecology who have achieved less than 2 years of their hole curriculum
  * Second group : trainees who have acieved at least 2 years and less than 4 years of the curriculum
  * third group : trainees who have achieved at least 4 years of their curriculum
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-30 (Estimated); Primary Completion 2022-01-03 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of surgical procedure needed for a trainee to master the FAUCS. | through study completion, an average of 1 year
  Number of surgical procedure needed for a trainee to acheive the highest evaluation

SECONDARY OUTCOMES:
operative time | through study completion, an average of 1 year
  time elapsed from skin incision and the end of surgery will be measured in minutes
neonatal acid base balance | immediately after birth
  cord blood gaz
new born overall condition | 5 minutes after birth
  Apgar score ( The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form an ackronym (Appearance, Pulse, Grimace, Activity, Respiration).he test is generally done at 1 and 5 minutes after birth and may be repeated later if the score is and remains low. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts .
calculated blood loss | the day and 24 hours after surgery
  changes in hematocrites levels before and after a surgery

CONTACTS AND LOCATIONS:
Overall Officials: kaouther dimassi, MD, Principal Investigator — University Tunis El Manar , Faculty of medicine Tunis
Locations (1):
- Kaouther Dimassi, Tunis, Marsa, Tunisia

IPD SHARING:
Plan to Share IPD: No